CLINICAL TRIAL: NCT03707990
Title: A First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of Single Doses of NNC0165-1875 as Monotherapy and in Combination With Semaglutide in Subjects With Overweight or Obesity
Brief Title: A Research Study of NNC0165-1875 Alone or Together With Semaglutide in People Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9775-4398; U1111-1212-3615 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: In total, 11 cohorts are planned. Five cohorts in Part 1 (cohort 1-5), and 6 cohorts (cohort 6-11) in Part 2. Each cohort will contain 8 participants. The first 2 participants will be randomised so one participant will receive active (Part 1: NNC0165-1875; Part 2: NNC0165-1875 and semaglutide) while the other receive placebo (Part 1: placebo; Part 2: placebo and semaglutide) treatment. The participants will remain in-house for a 5 days safety observation period. The remaining 6 subjects will be dosed at least after 96 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0165-1875 (Experimental): Participants will receive NNC0165-1875 alone in cohorts 1-5 (part 1) and NNC0165-1875 along with semaglutide in cohorts 6-11 (part 2).
  Interventions: Drug: NNC0165-1875; Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo alone in cohorts 1-5 (part 1) and placebo along with semaglutide in cohorts 6-11 (part 2).
  Interventions: Drug: Placebo (NNC0165-1875); Drug: Semaglutide

INTERVENTIONS:
Drug: NNC0165-1875 — Participants will receive a single dose of subcutaneous (s.c.) NNC0165-1875 injection. The planned doses of NNC0165-1875 are as following: cohort 1 and 7: 0.1 mg, cohort 2 and 8: 0.3 mg, cohort 3 and 9: 0.6 mg, cohort 4 and 10: 1.2 mg, cohort 5 and 11: 2.4 mg and cohort 6: 0.03 mg.
  Arms: NNC0165-1875
Drug: Placebo (NNC0165-1875) — Participants will receive a single dose of s.c. placebo injection.
  Arms: Placebo
Drug: Semaglutide — Participants will receive a single dose of s.c. semaglutide 0.25 mg injection.

SUMMARY:
The study is looking at possible new medicines for weight control in people with high body weight. The study looks at how the new medicines work in the body. The study consists of two parts. If participants take part in Part 1, they will either get a single dose of NNC0165-1875 or a "dummy" medicine (placebo). If participants take part in Part 2, they will either get a single dose of NNC0165-1875 or "dummy" medicine and also a single dose of semaglutide. Which treatment participants get is decided by chance. For Part 1 participants will get 1 injection. For Part 2 participants will get 2 injections. A study nurse at the clinic will inject the medicine with a thin needle in a skin fold in the stomach. The study will last for about 9 weeks. Participants will have 7 visits to the clinic with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator
* Body weight greater than or equal to 70 kg

Exclusion Criteria:

- Male of reproductive age who or whose partner(s) is not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | Day 1-36
  Count of adverse events.

SECONDARY OUTCOMES:
AUC0-∞,1875,SD; the area under the NNC0165-1875 plasma concentration-time curve from time 0 to infinity after a single s.c. dose | 1-36 days
  Calculated based on plasma NNC0165-1875 measured (nmol*h/L) in blood.
Cmax,1875,SD; the maximum plasma concentration of NNC0165-1875 after a single s.c. dose | 1-36 days
  Calculated based on plasma NNC0165-1875 measured (nmol/L) in blood.
AUC0-∞,sema,SD; the area under the semaglutide plasma concentration-time curve from time 0 to infinity after a single s.c. dose | 1-36 days
  Calculated based on plasma semaglutide measured (nmol*h/L) in blood.
Cmax,sema,SD; the maximum plasma concentration of semaglutide after a single s.c. dose | 1-36 days
  Calculated based on plasma semaglutide measured (nmol/L) in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results